CLINICAL TRIAL: NCT00714532
Title: A Stage-Based Scheduled Smoking Intervention for Chinese
Brief Title: Smoking Reduction and Cessation Interventions for Chinese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California (Other)
Responsible Party: Principal Investigator, Janice Tsoh, Ph.D., Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14RT-0160H; TRDRP grant: 14RT-0160H; H10315-27252-03B
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; Asian American; Chinese American; smoking reduction; stage-based intervention; expert system; nicotine replacement; counseling
MeSH Terms: conditions — Smoking Cessation; Smoking Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Expert system only, which includes a stage-matched manual, and a series of 3 individualized tailored feedback reports at baseline, 1, and 3 months.
  Interventions: Behavioral: Expert System Only
- 2 (Experimental): The intervention consists of 3 components:
  * Expert system which includes a stage-matched manual, and a series of 3 individualized tailored feedback reports at baseline, 1, and 3 months
  * scheduled smoking intervention, which includes a tailored-made 3-week smoking reduction schedule and a stage-matched tip guide to explain why and how to use the smoking reduction intervention
  * telephone check-in calls to provide brief counseling and technical support to motivate participants to use the intervention materials
  * a 2-week supply of nicotine gum or lozenge per participants' choice to use during smoking reduction
  Interventions: Behavioral: Enhanced Expert System

INTERVENTIONS:
Behavioral: Expert System Only — Expert system which includes a stage-matched manual, and a series of 3 individualized tailored feedback reports at baseline, 1, and 3 months
  Arms: 1
Behavioral: Enhanced Expert System — The intervention consists of 3 components:
  * Expert system which includes a stage-matched manual, and a series of 3 individualized tailored feedback reports at baseline, 1, and 3 months
  * scheduled smoking intervention, which includes a tailored-made 3-week smoking reduction schedule and a stage-matched tip guide to explain why and how to use the smoking reduction intervention
  * telephone check-in calls to provide brief counseling and technical support to motivate participants to use the intervention materials
  * a 2-week supply of nicotine gum or lozenge per participants' choice to use during smoking reduction
  Arms: 2

SUMMARY:
This study aims at developing and testing a stage-based scheduled smoking intervention that targets to encourage smokers to reduce smoking and to facilitate smoking abstinence. We hypothesize that smokers who receive the staged-based scheduled smoking intervention will be more likely to report smoking abstinence, quit attempts, and smoking reduction at 12 months.

DETAILED DESCRIPTION:
The objective of the study is to document and systematically investigate the use of smoking reduction and cessation strategies targeting Chinese American smokers at various level of readiness to quit smoking.

Using a randomized controlled study design, the experimental intervention will be compared to a control group that will receive the expert system intervention only at 3-, 6- and 12-month follow-up. The primary aim is to test the following hypotheses:

1. Participants receiving the experimental intervention will be more likely to achieve at least a 50% reduction from baseline at 3-month (end of treatment), 6- and 12-month follow-up than participants in the control condition.
2. Participants receiving the experimental intervention will be more likely to report a 24- hour quit attempt at 3-, 6- and 12-month follow-up.
3. Participants receiving the experimental intervention will be report a longer length of abstinence in their quit attempts at 3-, 6- and 12-month follow-up.
4. The experimental condition will yield a higher rate of smoking abstinence at 3-, 6- and 12-month follow-up.

The secondary aim is to examine the feasibility of the proposed intervention which will be assessed by recruitment efficiency, refusal rates, adherence, usage, safety data, and perceived helpfulness of the intervention components. In addition, analyses will be pursued to explore both short- and long-term maintenance of smoking reduction achieved, the association between smoking reduction and changes in self-efficacy of resisting from smoking, stage movements (changes in readiness for quitting), and the use of coping strategies for smoking at follow-ups. The study will provide important empirical data for developing effective smoking cessation strategies that are culturally and linguistically appropriate for the Chinese American population.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified ethnic Chinese men and women
* 18 years or older
* report smoking cigarettes daily with at least 5 cigarettes per day in the last 7 days
* reside in California
* be able to read written English or Chinese

Exclusion Criteria:

* Currently engaging in assisted smoking cessation efforts
* Have health conditions that have contraindications of using nicotine replacement treatment (NRT) such as pregnancy, within 6 months post MI, severe or unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
self-report 7-day smoking abstinence | 12 months

SECONDARY OUTCOMES:
self-report a 24-hour quit attempt | 12 months
50% or more reduction in smoking from baseline | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Janice Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Langley Porter, San Francisco, California, United States